CLINICAL TRIAL: NCT00579150
Title: Exenatide Pregnancy Registry - Type 2 Diabetes in Pregnancy
Acronym: Exenatide
Status: Terminated | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5550C00004; BCA401 (Other: INC Research)
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Birth Defects; Type 2 Diabetes; Preterm Birth
Keywords: Birth Defects; High Risk Pregnancy; Type 2 Diabetes
MeSH Terms: conditions — Congenital Abnormalities; Diabetes Mellitus, Type 2; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Exenatide: Exposure to any form of exenatide during pregnancy for treatment of type 2 diabetes. Patients also taking Insulin may be included, though only as part of a combination treatment.
- Non-exenatide group: Exposure to non-insulin antidiabetic medication not including exenatide for treatment of pre-existing type 2 diabetes during pregnancy. Patients also taking Insulin may be included, though only as part of a combination treatment.

SUMMARY:
This is an observational, prospective cohort study describing pregnancy outcomes in women with pre-existing (prior to pregnancy) type 2 diabetes who have been exposed to any formulation of exenatide during pregnancy. The pregnancy registry will compare the occurrence of the pregnancy outcomes of interest with those collected from a prospective group of women with pre-existing type 2 diabetes who have been exposed to one or more antidiabetic medications other than exenatide during pregnancy. Insulin exposures are acceptable in both groups but must be in addition to one or more other antidiabetic medications in the non-exenatide group.

The primary study objective is to evaluate the percentage of major birth defects (i.e., those that caused significant functional or cosmetic impairment, required surgery, or were life-limiting) following use of exenatide during pregnancy for treatment of type 2 diabetes compared to the percentage of major birth defects following use of one or more antidiabetic medications other than exenatide during pregnancy for treatment of type 2 diabetes.

The secondary objectives of the Exenatide Pregnancy Registry are to evaluate the percentage of other adverse pregnancy outcomes (e.g., spontaneous abortion, stillbirth, preterm birth) and any potential impact of exenatide use during breastfeeding among pregnancies or births in women who used exenatide for pre-existing type 2 diabetes:

This study is being conducted in the United States (US). Enrollment in the Registry is voluntary. The Exenatide Pregnancy Registry is sponsored by AstraZeneca and is managed by INC Research, LLC. The scientific conduct and analysis of the Registry is overseen by a Registry Review Committee (RRC) consisting of experts in maternal and fetal medicine, teratology/genetics, epidemiology, type 2 diabetes in pregnancy and/or pediatrics.

ELIGIBILITY:
Inclusion Criteria:

The subjects must meet the following eligibility criteria for participation in the registry:

* Is pregnant and at least 18 years of age at the time of enrollment
* Had a diagnosis of type 2 diabetes prior to pregnancy
* Does not know the pregnancy outcome at the time of enrollment
* Has no knowledge of any existing structural or chromosomal defects detected on a prenatal test prior to enrollment
* Had been exposed to an immediate release formulation of exenatide (e.g. BYETTA®) or a non-insulin antidiabetic medication other than exenatide on or after the first day of the last menstrual period (insulin use will be allowed for both groups). OR participant has been exposed to an extended release formulation of exenatide (e.g. BYDUREON®) within 8 weeks of the first day of the last menstrual period
* Is willing and able to provide informed consent and an authorization for the pregnancy registry to contact the obstetric HCP, diabetes HCP, and the infant's pediatric HCP (and complete contact information for these practitioners, if different, and if available)
* Is able to understand spoken English or Spanish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Is pregnant and at least 18 years of age at the time of enrollment
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2009-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | For each group, primary outcome measure will be assessed among all births, including major birth defects identified during the postnatal period and up to infant age 12 months.
  For each group, the primary outcome measure will be percentage of major birth defects-i.e., those that caused significant functional or cosmetic impairment, required surgery, or were life-limiting-among all births, including major birth defects identified during the postnatal period and up to infant age 12 months. For each group, the primary outcome measure will be percentage of major birth defects-i.e., those that caused significant functional or cosmetic impairment, required surgery, or were life-limiting-among all births, including major birth defects identified during the postnatal period and up to infant age 12 months.

SECONDARY OUTCOMES:
Secondary Outcome Measure | For each group, secondary outcome measures will be assessed among all identified pregnancies.
  For each group, the secondary outcome measure is to evaluate the percentage of the following outcomes among pregnancies or births in women with type 2 diabetes: Recognized spontaneous abortion (<20weeks gestation), Stillbirth (death of fetus at >/= weeks gestation, Preterm birth (<37 weeks gestation, infant macrosomia (>4,000 grams), low birth weight infants (<2,50o grams). To examine any potential impact of breastfeeding on infant growth during the first 4 months of life.

CONTACTS AND LOCATIONS:
Overall Officials: Vikki Brown, MD, Principal Investigator — Syneos Health; Esther Pascual, Study Director — AstraZeneca
Locations (1):
- Research Site, Wilmington, North Carolina, United States